CLINICAL TRIAL: NCT01073228
Title: A Randomized, Double-blind, Placebo-Controlled, Parallel, 24-Week, Phase 2 Study of Three Different Doses of an Alpha-7 Nicotinic Acetylcholine Receptor Agonist (EVP-6124) or Placebo in Subjects With Mild to Moderate Probable Alzheimer's Disease
Brief Title: Safety and Cognitive Function Study of EVP-6124 in Patients With Mild to Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: FORUM Pharmaceuticals Inc (Industry)
Collaborators: INC Research Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EVP-6124-010
Record Dates: First submitted 2010-02-19; First posted 2010-02-23 (Estimated); Last update posted 2014-04-25 (Estimated); Status verified 2013-02

CONDITIONS: Alzheimer's Disease; Central Nervous System Diseases; Cognition
Keywords: Alzheimer's disease; Central Nervous System diseases; Cognition
MeSH Terms: conditions — Alzheimer Disease; Central Nervous System Diseases | interventions — 7-chloro-N-quinuclidin-3-yl-benzo(b)thiophene-2-carboxamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- EVP-6124 0.3 mg (Active Comparator): one 0.3 mg capsule every day for 183 days
  Interventions: Drug: EVP-6124
- EVP-6124 1 mg (Active Comparator): one 1 mg capsule every day for 183 days
  Interventions: Drug: EVP-6124
- EVP-6124 2 mg (Active Comparator): one 2 mg capsule every day for 183 days
  Interventions: Drug: EVP-6124
- Placebo (Placebo Comparator): Placebo every day for 183 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EVP-6124
  Arms: EVP-6124 0.3 mg; EVP-6124 1 mg; EVP-6124 2 mg
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study is being conducted to determine the safety and effect on cognitive function of the investigational medication, EVP-6124, in individuals with mild to moderate probable Alzheimer's disease.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, parallel, 24-week, Phase 2 safety/efficacy study in which three dose levels of EVP-6124 or placebo will be evaluated. Eligible for enrollment will be patients who meet clinical criteria for mild to moderate probable Alzheimer's disease who are either receiving treatment with AChEI medication at a stable dose or who are not presently taking any AChEI or memantine co-medication.

Patients will be randomized to one of the following groups: 0.3 mg, 1 mg or 2 mg or Placebo. Approximately 400 subjects will be randomized to the 4 treatment groups. Study drug will be supplied as capsules and will be orally administered once daily for a total of 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with Probable Alzheimer's disease
* Mini-Mental State Examination (MMSE) score of 14 to 24 inclusive at screening and a CDR-SB score ≥2 at the screening assessment
* Modified Hachinski Ischemic Score (mHIS) ≤4 at screening
* Female subjects are ≥1 year post-menopausal or are surgically sterile
* Caregiver available; if not living in the same household, caregiver sees subject at least four times each week
* Subject living at home, senior residential setting, or an institutional setting without the need for continuous nursing care
* General health status acceptable for participation in a 24 week clinical trial be administered

Exclusion Criteria:

General

* Participation in another therapeutic clinical trial within 30 days before Baseline
* Prior participation in an amyloid vaccination clinical study
* Inability to swallow capsules
* Likely inability to complete 24 week study
* Inability to be ≥75% compliant with single-blind placebo run-in medication
* Inability to adequately perform cognitive tests
* History of significant cardiovascular disease
* Major depression
* Psychosis
* History of stroke within 18 months of screening
* Head trauma
* Inability to perform any screening or baseline evaluations

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 409 (Actual)
Dates: Start 2010-04; Primary Completion 2011-11 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Alzheimer's Disease Assessment Scale-Cognitive subscale-13 (ADAS-cog-13) | Day -7, Baseline, 4, 12, 18, 23 Weeks

SECONDARY OUTCOMES:
Alzheimer's Disease Assessment Scale-Cognitive subscale-11 | 4, 12, 18, 23 Weeks
Controlled Oral Word Association Test | Day -7, Baseline, 4, 12, 18, 23 Weeks
Category Fluency Test | Day -7, Baseline, 4, 12, 18, 23 Weeks
Clinical Dementia Rating Scale Sum of Boxes | Day -7, Baseline, 4, 12, 18, 23 Weeks
Alzheimer's Disease Cooperative Study-Activities of Daily Living | Baseline, 4, 12, 18, 23 Weeks
Neuropsychiatric Inventory | Baseline, 12, 23 Weeks
Mini-Mental State Exam | Day -7, Baseline, 4, 12, 18, 23 Weeks

CONTACTS AND LOCATIONS:
Locations (54):
- United States (25):
  - HOPE Research Institute, Phoenix, Arizona
  - Catalina Research Institute, Chino, California
  - ATP Clinical Research, Costa Mesa, California
  - University of California, Irvine, Orange, California
  - Radiant Research, Santa Rosa, California
  - Research Center for Clinical Studies, Inc., Norwalk, Connecticut
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - Meridien Research, Brooksville, Florida
  - Brain Matters Research, Delray Beach, Florida
  - MD Clinical, Hallandale, Florida
  - Galiz Research, Miami Springs, Florida
  - Renstar Medical Research, Ocala, Florida
  - Compass Research, LLC, Orlando, Florida
  - Princeton Medical Institute, Princeton, New Jersey
  - Memory Enhancement Center of NJ, Toms River, New Jersey
  - Brooklyn Medical Institute, Brooklyn, New York
  - Social Psychiatry Research Institute, Brooklyn, New York
  - Advanced Bio Behavioral Sciences Inc., Elmsford, New York
  - University of Rochester Medical Center at MCH, Rochester, New York
  - Columbus Research and Wellness Institute, Columbus, Ohio
  - Summit Research Network, Portland, Oregon
  - FutureSearch Trials of Dallas, L.P., Dallas, Texas
  - Grayline Clinical Drug Trials, Wichita Falls, Texas
  - The Memory Clinic, Bennington, Vermont
  - The Center for Excellence in Aging and Geriatric Health, Williamsburg, Virginia
- Romania (8):
  - Clinical Site 1, Bucharest
  - Clinical Site 2, Bucharest
  - Clinical Site 3, Bucharest
  - Clinical Site 4, Bucharest
  - Clinical Site 5, Bucharest
  - Iași
  - Oradea
  - Târgu Mureş
- Russia (10):
  - Kazan'
  - Clinical Site 1, Moscow
  - Clinical Site 2, Moscow
  - Clinical Site 1, Saint Petersburg
  - Clinical Site 2, Saint Petersburg
  - Clinical Site 3, Saint Petersburg
  - Clinical Site 4, Saint Petersburg
  - Saratov
  - Voronezh
  - Yekaterinburg
- Serbia (4):
  - Clinical site 1, Belgrade
  - Clinical Site 2, Belgrade
  - Kragujevac
  - Niš
- Ukraine (7):
  - Dnipro
  - Donets'k
  - (1), Kyiv
  - (2), Kyiv
  - Odesa
  - Simferopol
  - Vinnytsia